CLINICAL TRIAL: NCT01862731
Title: Vasti Control of Patellofemoral Kinematics in Patients With Chronic Patellofemoral Pain.
Brief Title: Muscle Strength Loss and Its Effect on Knee Cap Motion in Volunteers With Anterior Knee Pain
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 130099; 13-CC-0099
Record Dates: First submitted 2013-05-23; First posted 2013-05-24 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-12-10

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Muscle Force; Knee; Magnetic Resonance Imaging; Quadriceps; Ultrasound; Natural History
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Control Volunteers: Healthy controls
- 2/Volunteers with Pain: Subjects with Chronic Idiopathic Patellofemoral Pain

SUMMARY:
Background:

- Researchers are interested in how the muscles affect the movement of the knee cap. These muscles may be related to different kinds of knee pain that are not caused by an injury or a disease. Imaging studies such as magnetic resonance imaging (MRI) can be used to look at these muscles. To study these muscles and how they move, researchers will use MRI to look at healthy individuals and individuals with knee cap pain.

Objectives:

- To study how changes to the muscles around the knee can influence knee pain.

Eligibility:

* Individuals between 18 to 55 years of age who have knee cap pain that cannot be explained by a specific injury or disease.
* Healthy volunteers between 18 and 55 years of age.

Design:

* Participants will be screened with a physical exam and medical history.
* This study requires two visits. Each visit will use standard MRI sequences to take images of the knee in motion and at rest.
* On the first visit, the MRI scan will look at the knee in its natural state. Participants will move the knee up and down for 1 to 3 minutes at a time during the scan.
* On the second visit, a local anesthetic agent will be injected into the muscle of the thigh. The anesthetic will block this muscle from generating force for 2 or 3 hours. Participants will move the knee up and down for 1 to 3 minutes at a time during the MRI scan.

DETAILED DESCRIPTION:
Chronic idiopathic patellofemoral pain, a potential precursor to osteoarthritis, is one of the most common problems of the knee. It is characterized by anterior knee pain that is aggravated by deep knee flexion, prolonged sitting, and repetitive flexion/extension. The most widely accepted theory in regards to the source of this pain is that a force imbalance around the knee leads to static patellofemoral malalignment and dynamic patellofemoral maltracking. In turn, this malalignment and maltracking leads to elevated joint contact stresses, which ultimately leads to patellofemoral pain. Current understanding of patellofemoral maltracking is typically focused on static 2D alignment (lateral tilt and displacement). Yet, patellofemoral pain is most often exacerbated during dynamic events and the patella has complete six degrees of freedom in its movement. More recent studies have been able to quantify patellofemoral kinematics during volitional dynamic tasks and demonstrate that the maltracking problem is more complex than originally postulated. Specifically, in patients with patellofemoral pain, altered kinematics are not limited to excessive patellar lateral translation and tilt, but include excessive patellar superior translation along with excessive flexion and valgus rotations. Flexion and valgus are sagittal and coronal plane rotations that cause the superior pole of the patella to shift anteriorly and medially, respectively. Recent work has shown that altered force balance around the knee can indeed lead to maltracking. However, the question remains whether correcting an existing force imbalance around the knee can normalize patellar kinematics and/or reduce pain. The purpose of this study is to determine how temporary iatrogenic loss of force in the vastus lateralis muscle alters the aberrant patellar kinematics in subjects with chronic idiopathic patellofemoral pain.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male and female volunteers between the ages of 18 and 55

EXCLUSION CRITERIA:

All Volunteers

1. Any relevant medical problems, including 933 those preventing ambulation
2. Any serious injury to the joint being studied, previous surgery on the joint being studiedor extreme pain at the joint being studied or other condition that may explain the presence of PF_pain (e.g., meniscal tear, arthritis)
3. Allergy/hypersensitivity to any local anesthetic agent (e.g., Novocain, lidocaine, bupivacaine, ropivacaine)
4. Liver disease
5. Open angle glaucoma
6. Cardiac arrhythmias, congenital heart disease
7. Glucose-6-phosphate dehydrogenase deficiency
8. Any female who is pregnant

A volunteer will be excluded if they have a contraindication to MR imaging. Examples are:

1. Metal within their body, which might be expected to concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field (e.g., aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker or autodefibrillator, cochlear implant, other foreign body (e.g. metal shavings, insulin pump).
2. A condition, which would preclude them from participating in an MR imaging study (e.g., paralyzed hemidiaphragm, morbid obesity, severe claustrophobia)
3. A condition that presents an unnecessary risk to them or their unborn child (e.g., 953 pregnancy, previous surgery of uncertain type, symptoms of pheochromocytoma or insulinoma)

Subjects with Chronic Idiopathic Patellofemoral Pai:

1. Lack of PF_pain (either no active pain or current pain of < 6 months duration)

Control Volunteers:

1. Any clinical signs of a knee impairment in the joint being studied, including abnormal range of motion, muscle weakness, malalignment, and ligament damage.
2. The presence of PF_pain (either active or past)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited primarily from the greater Washington DC area. It will be advertised through clinicaltrials.gov, social media, flyers, and word of mouth.@@@
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
PF kinematics and the level of pain experience by the subject | prior to and after a nerve block
  The change in patellofemoral kinematics, patellofemoral pain, and quadriceps strength pre- and post-muscle block.

CONTACTS AND LOCATIONS:
Overall Officials: Frances T Gavelli, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
If other investigators wish to use these data, IRB approval will be sought prior to any data sharing. Data sharing will be done under a waiver of informed consent if (1) the previously signed consent form lacked data sharing information or (2) the consent form contained this information and the participant did not ask that his/her data not be shared. Waiver of consent meets the criteria set out in 45 CFR 46.116(d): The research and data sharing involves no more than minimal risk to the subjects.@@@@@@The waiver or alteration will not adversely affect the rights and welfare of the subjects. Data and samples will have personally identifying information removed.@@@The research could not practicably be carried out without the waiver or alteration.@@@Whenever appropriate, the subjects will be provided with additional pertinent information after@@@participation.
Supporting Information: ICF
Time Frame: Data will be shared through data sharing agreements.@@@@@@@@@@@@The start and end date will be determined by the data sharing agreement.
Access Criteria: Data will be shared stripped of PII and with IRB approval.

REFERENCES:
- [Background] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Hootman JM, Helmick CG. Projections of US prevalence of arthritis and associated activity limitations. Arthritis Rheum. 2006 Jan;54(1):226-9. doi: 10.1002/art.21562. PMID 16385518
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-CC-0099.html